CLINICAL TRIAL: NCT02300597
Title: Internet-based Support and Coaching for Adolescents and Young Adults With ADHD and Autism Spectrum Disorders - a Controlled Study
Brief Title: Internet-based Support for Young People With ADHD and Autism - a Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Södra Älvsborg Hospital (Other); Habilitation Services in Skaraborg, Skövde (Other)
Responsible Party: Principal Investigator, Elisabet Wentz, Associate professor, Göteborg University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBSC-2
Record Dates: First submitted 2014-11-10; First posted 2014-11-25 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: ADHD; Autism Spectrum Disorders
Keywords: ADHD; Autism Spectrum Disorders; controlled; Internet based; coaching
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet based support and coaching (Experimental): Young people between age 15 and 25 with ADHD and/or autism spectrum disorders are offered internet-based support and coaching during eight weeks (chat and e-mail). Data is collected before and after the intervention and six months after end of treatment using self-report questionnaires pertaining to sense of coherence, self-esteem, quality of life, depressive and anxiety symptoms and socioeconomic status. Parents complete an assessment scale for the next of kin. After treatment the young people are interviewed regarding the quality of the intervention.
  Interventions: Other: Internet based support and coaching
- Treatment as usual (TAU) (No Intervention): A comparison group matched for age, gender and neuropsychiatric diagnosis is offered treatment as usual and is assessed at the same time points as the intervention group.

INTERVENTIONS:
Other: Internet based support and coaching — Young people between age 15 and 25 with ADHD and/or autism spectrum disorders are offered internet-based support and coaching during eight weeks (chat and e-mail). Data is collected before and after the intervention and six months after end of treatment using self-report questionnaires pertaining to sense of coherence, self-esteem, quality of life, depressive and anxiety symptoms and socioeconomic status. Parents complete an assessment scale for the next of kin. After treatment the young people are interviewed regarding the quality of the intervention.
  Arms: Internet based support and coaching

SUMMARY:
Young people between age 15 and 25 with ADHD and/or autism spectrum disorders are offered internet-based support and coaching during eight weeks (chat and e-mail). Data is collected before and after the intervention and six months after end of treatment using self-report questionnaires pertaining to sense of coherence, self-esteem, quality of life, depressive and anxiety symptoms and socioeconomic status. Parents complete an assessment scale for the next of kin. After treatment the young people are interviewed regarding the quality of the intervention. A comparison group matched for age, gender and neuropsychiatric diagnosis is offered treatment as usual and is assessed at the same time points as the intervention group. The individuals are not randomized due to difficulties to recruit if the individuals do not know group assignment in advance.

DETAILED DESCRIPTION:
Young people between age 15 and 25 with ADHD and/or autism spectrum disorders are consecutively included in the project and are offered coaching and support during eight weeks over the internet (chat and e-mail) twice a week. Data is collected before and after the intervention as well as six months after end of treatment using self-report questionnaires (Sense of Coherence (SOC), Rosenberg Self Esteem Scale, Manchester Short Assessment of Quality of Life (MANSA), Montgomery Asberg Depression Rating Scale (MADRS), and Hospital Anxiety and Depression Scale (HAD)). A parent or a partner completes an assessment scale for the next of kin. When treatment is completed, the young people are interviewed using a structured interview pertaining to the quality of the intervention. A comparison group matched for age, gender and neuropsychiatric diagnosis is offered treatment as usual (TAU) and is assessed at the same time points as the intervention group. The individuals are not randomized to the intervention and comparison groups due to difficulties to recruit if the individuals do not know group assignment in advance. In all, 24 individuals will be offered the intervention and 24 individuals will receive TAU.

ELIGIBILITY:
Inclusion Criteria:

* ADHD and/or autism spectrum disorder
* Age 15 to 30

Exclusion Criteria:

* No current antisocial behaviour, psychotic symptoms and/or alcohol/substance abuse

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2010-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
QoL | T2: immediately after intervention; T3: 6 months after intervention. Outcome Measure is going to report a change.
  Self report questionnaire; Manchester Short Assesment of Quality of Life (MANSA), Priebe et. al. 1999.

SECONDARY OUTCOMES:
Self esteem | T2: immediately after intervention; T3: 6 months after intervention
  Self report questionnaire; Rosenberg Self-Esteem Scale (Rosenberg, 1965, 1989)
Sense of coherence | T2: immediately after intervention; T3: 6 months after intervention
  Self report questionnaire; Sense of Coherence (SOC-29), Antonovsky, 1987.
Anxiety and depressive symptoms | T2: immediately after intervention; T3: 6 months after intervention
  Self report questionnaire; Hospital Anxiety and Depression Scale (HAD), Zigmond & Snaith, 1983.
Depressive symptoms | T2: immediately after intervention; T3: 6 months after intervention
  Self report questionnaire; Montgomery Asberg Depression Rating Scale (MADRS), Montgomery & Asberg, 1979.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Neurochemistry, Institute of Neurosceince and Physiology, Gothenburg, Sweden

REFERENCES:
- [Derived] Sehlin H, Hedman Ahlstrom B, Andersson G, Wentz E. Experiences of an internet-based support and coaching model for adolescents and young adults with ADHD and autism spectrum disorder -a qualitative study. BMC Psychiatry. 2018 Jan 18;18(1):15. doi: 10.1186/s12888-018-1599-9. PMID 29347983